CLINICAL TRIAL: NCT00568126
Title: A Double-Blind, Placebo Controlled Study of Maca Root for the Treatment of Antidepressant-Induced Sexual Dysfunction in Females
Brief Title: Study of Maca Root for the Treatment of Antidepressant-Induced Sexual Dysfunction in Females
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); A Healthy Alternative, LLC (Other)
Responsible Party: Principal Investigator, David Mischoulon, MD, PhD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007P001090; R21AT004385 (NIH)
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Antidepressant Induced Sexual Dysfunction
Keywords: Antidepressant Induced Sexual Dysfunction; Depression; Sexual Dysfunction
MeSH Terms: conditions — Depression; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Subjects were randomized in a double blind manner to maca root or placebo. Improvement in sexual functioning was compared between the two treatment groups.
Who Masked: Participant, Investigator
Masking Description: Study subjects and investigator clinicians were blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maca Root (Experimental): Subjects in this arm will be given 3g/day of maca root for 12 weeks
  Interventions: Drug: Maca Root
- Placebo (Placebo Comparator): Subjects in this arm will receive inactive placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maca Root — 3g/day of Maca Root for 12 weeks.
  Other Names: Lepidium
  Arms: Maca Root
Drug: Placebo — Placebo provided by research pharmacy daily for 12 weeks.
  Other Names: Inactive placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out whether Maca Root is effective for treating sexual dysfunction in females that is caused by antidepressant drugs. An additional aim of the study is to document the safety and tolerability of maca root, as well as any potential side effects that it causes.

DETAILED DESCRIPTION:
This is a 12-week, double-blind, placebo-controlled trial comparing maca root (3.0 g/day) versus an inactive placebo in female outpatients with SSRI/SNRI-induced sexual dysfunction whose depression had remitted with SSRI treatment. Outcome measures include improvement in sexual functioning as per the Arizona Sexual Experience Scale (ASEX) and the Massachusetts General Hospital Sexual Function Questionnaire (MGH-SFQ).

ELIGIBILITY:
Inclusion Criteria:

* Subject is female, age 18 to 80 years
* Subject has been taking an SSRI, venlafaxine, or tri/heterocyclic antidepressant for the treatment of depression for at least 8 weeks; and is currently on a stable dose of the antidepressant for at least 4 weeks
* Subject is currently euthymic (HAM-D < 10) and is without significant anxiety symptoms (HAM-A < 10)
* Subject must have had no sexual dysfunction prior to taking antidepressant and there must be a clear temporal relationship between the sexual dysfunction and the antidepressant treatment
* Subject must have been consistently experiencing at least one of the following criteria for at least 4 weeks, with distress or disability:

  * Inability to have an orgasm, according to patient opinion
  * Clinically significant orgasm delay with masturbation or intercourse
  * Inability to attain or maintain until completion of sexual activity an adequate lubrication swelling response of sexual excitement
  * Decreased libido according to patient opinion
* Subject must be having or had been having some form of regular sexual activity (masturbation, oral sex, intercourse) at least twice monthly prior to the antidepressant treatment and are willing to continue efforts at sexual activity at least once weekly for the duration of the study
* Subject must be in good general physical health
* Subject must be able to understand and communicate in English
* Subject must have given informed consent to participate in the study

Exclusion Criteria:

* Primary or prior diagnosis of a sexual disorder (other than the side effect of the bipolar medication or symptom of the bipolar disorder)
* Sexual dysfunction secondary to general underlying medical condition
* Penile, vaginal, clitoral or other sexual organ anatomical deformities
* Any uncontrolled psychiatric disorder
* Alcohol or substance abuse or dependence within the past six months
* Recent major relationship changes, disruption, or turmoil ongoing or anticipated which are unrelated to her sexual dysfunction
* Hamilton Depression and/or Anxiety Scale score (either) > 10
* Blood pressure outside the range of 90/50 - 170/100
* Known hyperprolactinemia
* Use of investigational drugs within previous 3 months or during study
* Current use of other drugs for antidepressant induced sexual dysfunction or other therapies or medications to treat sexual dysfunction
* Current use of nefazodone
* Hormone replacement therapy, unless patient has been on stable dose of hormone therapy for at least 3 mo prior to the antidepressant treatment and had no sexual dysfunction while on the same hormone therapy regimen, and there is no change in the HRT during the study
* Pregnancy, lactating, or planning to become pregnant during the study
* Child bearing potential subjects unwilling and/or not prepared and/or who are judged unreliable to use an acceptable and verifiable form of contraception during the study
* Any clinically significant abnormality on the screening physical examination
* History of hormonal cancers
* Any medical or psychological condition or social circumstances that would impair subject's ability to participate reliably in the study, or that may increase the risk to subjects or others as a result of participating in this study
* Dyspareunia secondary to an inflammatory or anatomical condition
* Prior use of maca for at least two weeks
* Infection of the urogenital tract that may make sexual activity painful or difficult
* Subjects whose sexual partners are suffering from and/or receiving treatment for sexual dysfunction
* Receiving psychosexual or other therapy for sexual dysfunction and not willing to discontinue that treatment at screening
* Subjects who do not understand and communicate in English
* Subjects for whom sexual activity is inadvisable
* Subjects whose sexual dysfunction is considered to be situational
* Subjects not attempting some form of regular sexual activity at least twice monthly and at least once weekly during study visit intervals for duration of entire study
* Changes in antidepressant agent and/or dose of medication within the last 4 weeks before baseline visit
* Participants on medications with a narrow therapeutic window or low therapeutic index for which small variations may be harmful given the lack of systematic experience with drug-supplement interactions (i.e. - cyclosporine, digoxin, warfarin, and antiretrovirals)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-12-27 (Actual); Primary Completion 2010-10-05 (Actual); Study Completion 2010-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dording, MD, Principal Investigator — Massachusetts General Hospital; David Mischoulon, MD, PhD, Study Director — Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No current plan for this. In the event that other researchers inquire about using our data (e.g. in a meta-analysis), we will evaluate how to proceed.

REFERENCES:
- [Result] Dording CM, Schettler PJ, Dalton ED, Parkin SR, Walker RS, Fehling KB, Fava M, Mischoulon D. A double-blind placebo-controlled trial of maca root as treatment for antidepressant-induced sexual dysfunction in women. Evid Based Complement Alternat Med. 2015;2015:949036. doi: 10.1155/2015/949036. Epub 2015 Apr 14. PMID 25954318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study screened 57 and included 45 remitted depressed female outpatients aged 18-65. The patients were recruited from December of 2007 through June of 2010 through the Depression Clinical and Research Program in Boston, MA.
Pre-assignment Details: Patients were excluded if: diagnosed with a past sexual disorder, currently receiving other treatment for sexual dysfunction, experiencing sexual dysfunction due to underlying medical condition, had recent relationship changes or turmoil unrelated to the sexual dysfunction, or other health or social problems that might influence sexual dysfunction.
Period: Overall Study
Arm/Group | Maca Root | Placebo
Started | 24 | 21
Completed | 13 | 12
Not Completed | 11 | 9
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 4 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Population: This study recruited 45 remitted depressed female outpatients aged 18-65 who were currently suffering from antidepressant induced sexual dysfunction, and whose depression was in remission.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maca Root | Placebo | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants in Remission Based on Arizona Sexual Experience Scale (ASEX) Score of 10 or Less After 12 Weeks of Treatment.
Description: Arizona Sexual Experience Scale (ASEX) consists of five items rating sexual drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm.The range of total score is 5-30 with the higher scores indicating greater sexual dysfunction. A total final score of 10 or less is considered to indicate remission of sexual dysfunction.
Time Frame: 12 weeks
Population: Analysis of 42 women who completed at least one clinical assessment after a minimum of seven days of treatment. This included 21 women (14 premenopausal and 7 postmenopausal) randomized to treatment with maca and 21 women (16 premenopausal and 5 postmenopausal) randomized to placebo.
Measure: Number; unit: participants
Arm/Group | Maca Root | Placebo
Number analyzed (Participants) | 21 | 21
participants | 2 | 1
Statistical Analysis 1: Comparison: Maca Root vs Placebo; Treatment groups were compared based on percentage reaching remission thresholds per scale: a total score of 12 ("minimally diminished") or less on the MGH-SFQ scale, and a total score of 10 ("very strong/very easily/very satisfying") or less on the ASEX; Test type: Superiority — Remission rates for maca vs. placebo were compared by chi-squared and by odds ratio (with 95% confidence interval); p = 0.55, Chi-squared — P values above are calculated. No multiple comparisons. Threshold for significance set a priori as P<0.05; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.18 to 25.2] — Odds ratio for attaining remission while taking maca vs taking placebo

2. Primary Outcome: Proportion of Participants in Remission Based on Massachusetts General Hospital Sexual Functioning Questionnaire (MGH-SFQ) Score of 12 or Less After 12 Weeks of Treatment.
Description: Massachusetts General Hospital-Sexual Functioning Questionnaire (MGH-SFQ) is composed of five items evaluating libido, sexual arousal or excitement, ability to achieve orgasm, ability to achieve and maintain an erection (for men only) and overall sexual satisfaction. Items are rated on a scale of 1 to 6 with a rating of 1 indicating greater than normal functioning and a rating of 6 indicating totally absent functioning. A total final score of 12 or less is considered to indicate remission of sexual dysfunction.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Maca Root | Placebo
Number analyzed (Participants) | 21 | 21
participants | 6 | 4
Statistical Analysis 1: Comparison: Maca Root vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Remission rates for maca vs. placebo were compared by chi-squared and by odds ratio (with 95% confidence interval); p = 0.47, Chi-squared — P values above are calculated. No multiple comparisons. Threshold for significance set a priori as P<0.05; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.40 to 7.34] — Odds ratio for attaining remission while taking maca vs taking placebo

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from each patient over 12 weeks of treatment.
Description: Adverse events were recorded by study clinicians in the chart at each biweekly treatment visit over the 12-week course of treatment. The overall duration of the study was from December of 2007 through September of 2010 (2 years and 9 months).
Arm/Group | Maca Root | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 17/24 | 5/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maca Root (N=24) | Placebo (N=21)
Acute Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Increased appetite (Gastrointestinal disorders) | 3 (3) | 0 (0)
Weight Gain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 2 (2) | 2 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
1. Small sample. Reliance on patient self-report in domain of orgasm (subjective and subject to bias/inaccuracy). 2. No liver function tests (LFTs) obtained; some herbal extracts may induce LFT elevation, though there is no such evidence for maca.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No